CLINICAL TRIAL: NCT06591897
Title: Exploration of Gender Differences in Liver Aging
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0815
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Healthy Population
Keywords: hepatocyte; liver function; sex differences

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue of segment IV ( about 1mm³ )
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The liver is an important metabolic organ in the body. It participates in central metabolic activities to maintain systemic homeostasis. It is also one of the most vulnerable organs in the process of individual aging. During aging, the volume, blood flow, metabolic capacity and regenerative capacity of the liver decrease. Liver function changes with age can lead to age-related systemic susceptibility diseases.

Therefore, understanding the changes of metabolism and immune function in the process of liver aging and studying the regulation mechanism of liver aging will provide an important reference for understanding the causes of increased susceptibility to liver-related diseases in the elderly population.On the other hand, gender factors also affect organ function, leading to differences in human aging and disease outcomes.At present, the omics research on liver aging is mainly based on tissue-level transcription, protein or metabolomics, and most of the conclusions are focused on hepatocytes. However, for other cell types and microenvironment interactions, people know little about the aging changes at the cellular levelBased on the current research status, this study aims to explore the gender differences in the process of liver aging, using emerging technologies such as the combination of single-cell multi-omics and spatial localization, to reveal the factors driving liver aging from a gender perspective, and to promote the development of accurate interventions for aging and aging-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Liver function indicators are in the normal reference range.
* Liver imaging examination showed normal.

Exclusion Criteria:

* Patients with previous liver-related diseases.
* Subjects with important organ dysfunction / failure or other serious diseases ( myocardial infarction, malignant tumor, severe neurological or psychiatric history, severe infection, coagulation dysfunction, etc. )
* Moderate malnutrition ( BMI < 17kg / m2 ) and severe anemia ( Hb < 60g / L ).
* Subjects and their families who disagreed with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, the normal liver sampling criteria are as follows : 1.Preoperative blood biochemical liver function indicators are in the normal reference range.
  2.Liver imaging is normal. The liver is normal in size, regular in shape, smooth in capsule, uniform in parenchymal echo, and intrahepatic vascular network.
  For patients undergoing laparoscopic cholecystectomy, the liver tissue of the IV segment of the liver ( about 1mm3 ) was separated from the gallbladder wall specimen.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Molecular and cellular characteristics during liver aging | 2027.08
  Draw the map information of liver aging single cell precision, and clarify whether the effect of aging on liver cell types has gender differences.

CONTACTS AND LOCATIONS:
Overall Officials: daren Liu, MD, PhD, Study Director — Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No